CLINICAL TRIAL: NCT03343548
Title: The Effect of Adjuvant Epidural Magnesium Sulfate to Bupivacaine and Morphine on Post-thoracotomy Pain Control: A Randomized Double Blind Clinical Trial Study
Brief Title: Epidural Magnesium Sulfate for Post-thoracotomy Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Institute of Tuberculosis and Lung Disease, Iran (Other Government)
Responsible Party: Principal Investigator, Shadi Baniasadi, Dr, National Research Institute of Tuberculosis and Lung Disease, Iran
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1019-211194
Record Dates: First submitted 2017-11-12; First posted 2017-11-17 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): magnesium group (Mg)
  Interventions: Drug: magnesium sulfate
- Group II (Placebo Comparator): control group (C)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: magnesium sulfate — 2cc of magnesium sulfate ( 50%) will be administered epidurally
  Arms: Group I
Drug: normal saline — 2cc of normal saline will be administered epidurally
  Arms: Group II

SUMMARY:
Pain after thoracotomy is very severe and may cause pulmonary complications. Thoracic epidural analgesia has greatly decreased the pain experience and its consequences. However, new ways of decreasing post-operative opioid drugs consumption is an important issue of research. We aim to evaluate the effect of adding epidural magnesium sulfate to bupivacaine and morphine on pain control and the amount of opioid consumption after thoracotomy. Eighty patients undergoing thoracotomy at a tertiary cardiothoracic referral center will be enrolled in a randomized double blind trial. Patients randomly will be allocated in two groups. Bupivacaine (12.5 mg) plus morphine (2 mg) will be administered epidurally for all patients at the end of operation. Patients in group I will be received epidural magnesium sulfate (50 mg) and patients in Group II will be received normal saline as an adjuvant. Visual analog scale (VAS) score and the amount of morphine consumption will be measured during 24 hours post-operation.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical statuses I-III
* Undergoing thoracotomy

Exclusion Criteria:

* Known hypersensitivity to magnesium sulfate
* Renal failure
* Hepatic dysfunction
* Severe obesity
* Psychotic or neurologic diseases
* Currently taking opioid or calcium channel blocker
* AV block degree II or III
* Refused to participate in trial

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
severity of post-thoracotomy pain | 24 hours after thoracotomy
  VAS (visual analog scale: 0-10 cm (0 cm = no pain and 10 cm = the worst pain)) score will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Shadi Baniasadi, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No